CLINICAL TRIAL: NCT02187484
Title: BIBR 277 Capsules Clinical Study on Hypertension With Nephropathy
Brief Title: BIBR 277 Capsules in Hypertensive Patients With Nephropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 502.266
Record Dates: First submitted 2014-07-09; First posted 2014-07-11 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2014-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan

ARMS (1):
- Single rising doses of BIBR 277 (Experimental)
  Interventions: Drug: BIBR 277

INTERVENTIONS:
Drug: BIBR 277

SUMMARY:
The antihypertensive effect, safety and usefulness of treatment with BIBR 277 capsules were evaluated in hypertensive patients with nephropathy

ELIGIBILITY:
Inclusion Criteria:

* Condition: Either of the following criteria is satisfied in laboratory tests:

  * Presence of a renal parenchymal disorder such as chronic glomerulonephritis is confirmed (serum creatinine < 3.0 mg/dL)
  * Presence of a renal function disorder (serum creatinine ≥ 1.5 mg/dL to < 3.0 mg/dL)
* Age: ≥ 20 years
* Sex: Either male or female
* Patient status: Either outpatients or inpatients. However, the patient status should remain unchanged throughout the study period
* Blood pressure (BP):

  * [Outpatients] The last 2 measurements of sitting BP out of at least 3 taken during the observation period (2 - 4 weeks) should be stable and a mean of the two measurements should be ≥160 mmHg for systolic BP (SBP) and ≥95 mmHg for diastolic BP (DBP)
  * [Inpatients] The last 2 measurements of supine BP taken during the observation period (1 week) should be stable and a mean of the 2 measurements should be ≥ 150 mmHg for SBP and ≥ 90 mmHg for DBP

Exclusion Criteria:

* Renovascular hypertension
* Undergoing haemodialysis
* Severe hypertension (Diastolic BP ≥ 120 mmHg)
* Severe heart failure, angina pectoris, or history of myocardial infarction
* Atrioventricular conduction disturbance (degree II to III), atrial fibrillation, or serious arrhythmia
* Symptoms of cerebrovascular disorder
* Serious hepatic dysfunction
* Uncontrolled diabetes
* Peptic ulcer
* History of hypersensitivity to drugs
* Hyperkalaemia
* Undergoing treatment with a digitalis preparation
* Pregnant, breast feeding, possibly pregnant or planning to become pregnant during this study
* Otherwise judged ineligible by the investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 1998-08; Primary Completion 1999-08 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in hypertensive effect by investigator, using a 5-grade classification | 8 weeks after start of treatment

SECONDARY OUTCOMES:
Changes from baseline in blood pressure reduction | 8 weeks after start of treatment
Rate of blood pressure normalisation | 8 weeks after start of treatment
  percentage of patients with < 150/90 mmHg
Changes from baseline in blood pressure / pulse rate | 8 weeks after start of treatment
Usefulness assessment by investigator, using a 5- grade classification | 8 weeks after start of treatment
Overall safety assessment by investigator, using a 5- grade classification | 8 weeks after start of treatment
Number of patients with adverse events | Up to 12 weeks
Number of patients with abnormal changes in laboratory values | Up to 8 weeks after start of treatment